CLINICAL TRIAL: NCT05631353
Title: Carriere Motion Appliance in The Treatment of Class II Malocclusion Using Different Methods of Anchorage Control (Cone Beam Study)
Brief Title: TADs Anchored vs Conventional Anchored Carriere Motion Appliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abdelshafy Ali, Assistant lecturer, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Carriere motion appliance
Record Dates: First submitted 2022-11-21; First posted 2022-11-30 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Class II Malocclusion
Keywords: Carriere Motion Appliance
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: data will be sent blinded for statistical analysis
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: Patients will be treated by Carriere Motion Appliance using passive lingual arch . (Active Comparator): Conventional mandibular anchorage During the first month, 1/4-inch heavy elastics will be used. In the following months, 3/16-inch heavy elastics will be used. The patients will be instructed to wear the elastics 24 hours per day, except during mealtimes, and to change them daily
  Interventions: Device: Carriere Motion Appliance
- Group II: Patients will be treated by Carriere Motion Appliance using direct mini-screw. (Active Comparator): TADs mandibular anchorage. During the first month, 1/4-inch heavy elastics will be used. In the following months, 3/16-inch heavy elastics will be used. The patients will be instructed to wear the elastics 24 hours per day, except during mealtimes, and to change them daily
  Interventions: Device: Carriere Motion Appliance

INTERVENTIONS:
Device: Carriere Motion Appliance — Patient will be randomly allocated into two groups:
  Group I: conventional mandibular anchorage using passive lingual arch. Group II: anchorage by direct mini-screws. In the group I, Class II elastics will be attached from the maxillary canine to the mandibular first molar bilaterally with passive lingual arch in the lower arch as anchorage means.
  In the group I, Class II elastics will be attached from the maxillary canine to mandiular miniscrews bilaterally.
  For each patient, two CBCT radiographs will be obtained: one preoperatively and another after completion of distalization.
  Other Names: Passive lingual arch.; Mini-screw.

SUMMARY:
Carriere Motion appliance (CMA) was designed to correct a Class II molar relationship into a Class I relationship by distalizing the whole posterior maxillary segment by means of class II elastics and mandibular anchorage. To revoke the adverse effects of CMA with class II elastics, we can use the CMA to distalize the maxillary posterior segment with TADs anchorage using miniscrews. The aim of this study is to evaluate TADs anchored CMA vs. conventionally anchored CMA for distalization of the maxillary buccal segment.

DETAILED DESCRIPTION:
Twenty class II malocclusion patients with age (11-16) years will be randomly allocated in the two groups:

Group I: Patients will be treated by Carriere Motion Appliance using passive lingual arch.

Group II: Patients will be treated by Carriere Motion Appliance using direct mini-screw.

For each patient, two CBCT will be obtained: one preoperatively and another after completion of distalization.

Comparing skeletal and dental measurements obtained from CBCT radiographs obtained prior to treatment (T0) and immediately after correction of class II and remval of the appliance (T1).

ELIGIBILITY:
Inclusion Criteria:

* Adolescent patients aged 11-17 years.
* Unilateral or bilateral Class II molar relationship.
* Bilateral Class II canine relationship.
* No history of previous orthodontic treatment.
* No malformed teeth, impacted teeth and unerupted teeth.
* No systemic disease.
* Good oral hygiene.
* No abnormal pressure habit.
* No periodontal diseases.
* No missing teeth in maxillary arch.

Exclusion Criteria:

* The need for extraction in the lower arch.
* Posterior crossbite.
* Presence of any craniofacial anomalies.
* Patients with syndromes.

Ages: 11 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-01 (Actual)

PRIMARY OUTCOMES:
Treatment duration | from date of appliance delivery to date of removal after reaching class I molar relationship (about 4-6 months)
  months
Skeletal changes | from date of appliance delivery to date of removal after reaching class I molar relationship (about 4-6 months) ]
  degrees
Dental changes | from date of appliance delivery to date of removal after reaching class I molar relationship (about 4-6 months)
  degrees

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Anwar El-sayed, professor, Study Chair — saleh.anwar@azhar.edu.eg
Locations (1):
- Alazhar university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Carriere L. A new Class II distalizer. J Clin Orthod. 2004 Apr;38(4):224-31. No abstract available. PMID 15115896
- [Background] Rodriguez HL. Unilateral application of the Carriere Distalizer. J Clin Orthod. 2011 Mar;45(3):177-80. No abstract available. PMID 21785202
- [Background] Wilson B, Konstantoni N, Kim KB, Foley P, Ueno H. Three-dimensional cone-beam computed tomography comparison of shorty and standard Class II Carriere Motion appliance. Angle Orthod. 2021 Jul 1;91(4):423-432. doi: 10.2319/041320-295.1. PMID 33560300